CLINICAL TRIAL: NCT01846104
Title: Safety and Immunogenicity of a Booster Dose (50 µg) of Recombinant Ricin Toxin A-Chain 1-33/44-198 (rRTA 1-33/44-198) Vaccine (RVEc™) in Previously Vaccinated Healthy Adults
Brief Title: Booster Dose (50 µg) of Recombinant Ricin Toxin Vaccine (RVEc™) in Previously Vaccinated Healthy Adults
Acronym: RVEc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-12-23; FY12-16 (Other: USAMRIID)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Ricin Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50-μg booster dose RVEc (Experimental): Subjects will be receive one 50-μg dose of RVEc
  Interventions: Biological: 50-μg booster dose RVEc

INTERVENTIONS:
Biological: 50-μg booster dose RVEc — Subjects will be recruited from the 10 subjects who received three 50-μg doses of RVEc during the Phase 1 trial. Subjects will receive a single booster dose only and will be followed for 6 months after vaccination.
  Other Names: Ricin Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single 50-μg booster dose of RVEc. Subjects will be recruited from the cohort that received three 50-μg doses of RVEc in a Phase 1 trial (NCT01317667).

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must have received the 3 priming doses of RVEc at the 50-µg dosage.
* Study subjects must be 18 years old at time of screening and no older than 50 years old at time of vaccination.
* Subjects must weigh at least 110 pounds at time of screening.
* Subjects must be in good health as judged from medical history, physical examination, EKG, hematology, clinical chemistries, urinalysis, hepatitis serology, and HIV antibody test (Table 4) and be medically cleared for participation by an investigator. If any HIV or hepatitis testing is positive, the individual will be provided with counseling and referral for health care.
* Females of child-bearing potential must have a negative pregnancy test on screening and the morning of vaccination prior to receipt of the vaccine and must agree to use a highly effective method of birth control during the first 3 months following receipt of RVEc. A highly effective method of birth control is defined as one with a failure rate of less than 1% per year. Acceptable birth control methods that meet this criterion include hormonal implants and injectables (Norplant, Depo-Provera, Lunelle, and Etonogestrel), combined oral contraceptives, the intrauterine devices (IUDs) Copper T (380-A) or Mirena (Levonorgestrel Intrauterine System), female sterilization (tubal ligation), sexual abstinence, or a vasectomized partner.
* Female subjects must also agree not to breastfeed until at least 3 months after receiving the RVEc.
* Study subjects must read and sign an approved informed consent.
* Study subjects must be willing to return for all follow-up visits.
* Study subjects must agree to report any AE that may or may not be associated with administration of the investigational product through the 6-month follow-up/closeout visit.
* Study subjects must agree to abstain from excessive exercise (more than the usual routine) and excessive alcohol consumption (exceeds more than 2 drinks for males or 1 drink for females daily or binge drinking) for the duration of study participation.

Exclusion Criteria:

* Acute or chronic medical conditions or immunodeficiency from a medical condition or medical treatment, medications, or dietary supplements that, in the investigator's opinion, would impair the subject's ability to respond to vaccination. Use of corticosteroids, other than inhaled corticosteroids, will not be permitted.
* Severe hypersensitivity to any vaccine (anaphylaxis, angioedema, bronchospasm, or laryngospasm).
* History of asthma, chronic obstructive pulmonary disease, or other current/residual diseases of the lungs.
* Clinically significant abnormal laboratory tests.
* Current smoker.
* Any known allergies to sodium succinate, Tween-20 (a detergent), aluminum hydroxide, or kanamycin.
* Receipt of any vaccine or investigational product within 30 days before or after vaccination with RVEc.
* Receipt of RVEc is contraindicated based on SIRVA checklist/screening, as determined by PI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Chambers, MD, MPH, Principal Investigator — USAMRIID
Locations (1):
- Department of Clinical Research, USAMRIID, Frederick, Maryland, United States

REFERENCES:
- [Result] Pittman PR, Reisler RB, Lindsey CY, Guerena F, Rivard R, Clizbe DP, Chambers M, Norris S, Smith LA. Safety and immunogenicity of ricin vaccine, RVEc, in a Phase 1 clinical trial. Vaccine. 2015 Dec 16;33(51):7299-7306. doi: 10.1016/j.vaccine.2015.10.094. Epub 2015 Nov 3. PMID 26546259

RESULTS

PARTICIPANT FLOW:
Groups:
- 50-μg Booster Dose RVEc: Subjects will be receive one 50-μg dose of RVEc
  50-μg booster dose RVEc: Subjects will be recruited from the 10 subjects who received three 50-μg doses of RVEc during the Phase 1 trial (NCT01317667). Subjects will receive a single booster dose only and will be followed for 6 months after vaccination.
Period: Overall Study
Arm/Group | 50-μg Booster Dose RVEc
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 50-μg Booster Dose RVEc
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaccinated Participants Who Experienced Adverse Events by Nature and Severity.
Time Frame: Six months
Population: All statistical analysis of safety data was conducted using 4 subjects at every time point except Day 180 (for which there were 3 subjects).
Measure: Number; unit: participants
Arm/Group | 50-μg Booster Dose RVEc
Number analyzed (Participants) | 4
participants
  Vaccinated without symptoms | 0
  Vaccinated with any severity of local reaction | 3
  Vaccinated with mild systemic reactions | 3
  Vaccinated with moderate systemic reactions | 2
  Vaccinated with severe systemic reactions | 1
  Vaccinated with life-threating systemic reaction | 0
  Vaccinated that developed hypernatraemia | 3
  Vaccinated that developed injection site pain | 3

2. Secondary Outcome: Number of Subjects Who Developed Total ELISA IgG Titers (≥ 1:500)
Time Frame: Six months
Population: All statistical analysis of immunogenicity data was conducted using 4 subjects at every time point except Day 84 and 180 (for which there were 3 subjects).
Measure: Number; unit: Subjects with Total ELISA IgG (≥ 1:500)
Arm/Group | 50-μg Booster Dose RVEc
Number analyzed (Participants) | 4
Subjects with Total ELISA IgG (≥ 1:500)
  Day 0 | 0
  Day 1 | 1
  Day 3 | 1
  Day 7 | 3
  Day 14 | 4
  Day 28 | 4
  Day 42 | 4
  Day 56 | 4
  Day 84 | 3
  Day 180 | 3

3. Secondary Outcome: Number of Subjects Who Developed TNA Anti-ricin Toxin-neutralizing Antibody Titers (≥ 1:50)
Time Frame: Six months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | 50-μg Booster Dose RVEc
Number analyzed (Participants) | 4
participants
  Day 0 | 0
  Day 1 | 0
  Day 3 | 0
  Day 7 | 3
  Day 14 | 4
  Day 28 | 4
  Day 42 | 4
  Day 56 | 4
  Day 84 | 3
  Day 180 | 3

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | 50-μg Booster Dose RVEc
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50-μg Booster Dose RVEc (N=4)
Injection site pain (General disorders) | 3 (3)
Migrain (Nervous system disorders) | 1 (1)
Temporo-mandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hyper-natraemia (Metabolism and nutrition disorders) | 3 (3)
Blood creatine phosphor-kinase increased (Investigations) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1)
Blood urea increased (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Four subjects were enrolled and vaccinated. Three subject completed the study and one was withdrawn due to relocation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No